CLINICAL TRIAL: NCT03236077
Title: Increasing Exercise Enjoyment and Outcome Expectations Among Women With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Community Foundation of Greater Buffalo (Unknown)
Responsible Party: Principal Investigator, Lucia A Leone, Assistant Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1134041
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: obesity, women, exercise, physical activity,
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Immunoglobulin Fab Fragments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Fit and Fab

INTERVENTIONS:
Behavioral: Fit and Fab — participate in a targeted exercise program at the YMCA. Will include: Targeted exercise classes, Strength-training, Group support sessions
  Arms: Intervention

SUMMARY:
Despite decades of physical activity (PA) research on inactive, obese individuals, we have not successfully moved the needle on exercise participation in this population. A recent review aptly referred to PA recommendations among obese individuals as "the public health guideline that is (almost) entirely ignored"[1]. While we have previously had little understanding of why PA rates are so low in this population, Dr. Leone's research uncovered two possible explanations: (1) women with obesity are less likely to report enjoying exercise and (2) more likely than non-obese women to report exercising only when they are trying to lose weight. In order to affect change among obese women, we need interventions that not only address disparities in enjoyment and outcome expectations. Programs must also be practical and scalable; however, these types of evidence-based programs do not exist within the context that people generally exercise (e.g., community centers, gyms). We propose a novel approach to increasing exercise participation in this population by focusing on exercise enjoyment, increasing appreciation of the proximal benefits of PA rather than focusing on weight, and addressing changes to the exercise environment that make it conducive to this population. By delivering our intervention in partnership with the YMCA, we not only have the ability to make changes to a typical exercise context, but we also ensure that our findings can be used to help exercise-focused community organizations implement a scalable, research-tested program.

DETAILED DESCRIPTION:
This is a pilot intervention study with two groups: an intervention group (targeted exercise program for women with obesity and YMCA membership) and a control group (YMCA membership only). The targeted exercise program will be delivered by a YMCA and will be evaluated by our team. The majority of women who are recruited to this study will be randomized to receive the intervention or the control condition. However, we also have a small group of women who has been serving as our community advisory committee (CAC) that will also participate in the intervention classes and receive the membership. They will serve as pilot testers for our data collection methods and provide ongoing qualitative feedback on the intervention as part of their role in the CAC.

The study will take place in two phases at two different YMCAs (Ken-Ton and Independent Health) with approximately half of participants recruited for the first and the other half for the second.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-64
* BMI ≥ 30 (self-reported for initial screening and confirmed at informational session using direct measurement)
* Not currently participating in any regularly scheduled exercise (see definition in eligibility screener)
* Willing to come to the Ken-Ton YMCA 2-3x/week (Phase 1) or the Independent Health YMCA (Phase 2)

Exclusion Criteria:

* - Participants may not be pregnant or planning to become pregnant in the next 6 months
* Individuals with disabilities or health conditions that render them unable to participate in exercise or for whom exercise might be dangerous based on their answers to the Physical Activity Readiness Questionnaire or advisement form their physician

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
YMCA attendance | 3 motnhs
  YMCA attendance measured by swipes of member card

SECONDARY OUTCOMES:
MVPA | 3 months
  Minutes/week of moderate-to-vigorous exercise measured via accelerometer

OTHER OUTCOMES:
Exercise Enjoyment | 3 months
  Report greater enjoyment and acceptability of the exercise measured by the Physical Activity Enjoyment Scale (PACES)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided